CLINICAL TRIAL: NCT00671021
Title: Evaluation of Duration of Platelet Inhibition by Aspirin in a Standard 24-hour Interval Dosing Regimen
Brief Title: Duration of Platelet Inhibition by Aspirin
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Other Study IDs: C.E. 2007-05-42
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
Keywords: platelet aggregation; aspirin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Platelet Aggregation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients suffering from stable CAD, on chronic ASA therapy
  Interventions: Other: Platelet aggregation

INTERVENTIONS:
Other: Platelet aggregation — Platelet aggregation TxA2 formation

SUMMARY:
The well established importance of regular aspirin administration stands on firm grounds, as large meta-analyses have shown this therapy to significantly reduce the risk of death. However, not all patients benefit of aspirin administration to the same extent, thus high-lighting a sub-population of patients with inadequate platelet response to ASA. The mechanisms underlying reduced ASA efficacy remain elusive. A recent report has suggested that platelets, long believed to be incapable of de novo protein synthesis, may retain their ability to form the cyclooxygenase enzyme, once it has been inactivated by aspirin. This may explain the inefficacy of the drug to induce sustained platelet inhibition in certain patients.

The current study aims to evaluate, in patients suffering from stable coronary artery disease, the stability of platelet inhibition by aspirin during the normal once daily dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stable CAD, on chronic ASA therapy
* Patients willing to participate in the study and to sign the informed consent form

Exclusion Criteria:

* Acute coronary syndrome or revascularization in the last 3 months prior to enrolment
* Concurrent ingestion of nonsteroidal anti-inflammatory drugs (NSAIDs, including COX-2 selective anti-inflammatory drugs), clopidogrel, ticlopidine, dipyridamole, warfarin or acenocoumarol
* Frequent use (more than once a week) of non-prescription NSAIDs or drugs containing ASA in the 10 days preceding enrolment
* Major surgical procedure within 1 month before enrolment
* Hemorrhagic diathesis or known platelet dysfunction
* Platelet count outside the 100 to 450 x109/L range for technical reasons
* Hematocrit < 25% or haemoglobin < 100 g/L
* Patient undergoing dialysis for chronic renal failure
* Patient found to be ASA resistant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from stable CAD, on chronic ASA therapy
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation TxA2 formation

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Diodati, MD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada